CLINICAL TRIAL: NCT02676206
Title: Music Therapy in Procedural Sedation in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-540
Record Dates: First submitted 2016-01-28; First posted 2016-02-08 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2022-04

CONDITIONS: Conscious Sedation Failure During Procedure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music intervention (Experimental): Subjects will have headphones placed on 1 minute prior to procedural sedation. Classical music will be played until the subject is fully awake.
  Interventions: Other: Classical music
- Non intervention (No Intervention): Subjects will have headphones placed on 1 minute prior to procedural sedation. No music will be played. The headphones will be removed when the subject is fully awake.

INTERVENTIONS:
Other: Classical music — Classical music will be played over the headphones
  Other Names: Intervention arm
  Arms: Music intervention

SUMMARY:
The investigators propose to determine whether listening to classical music during a sedation procedure decreases the need for procedural sedation medication. It is a two arm study comparing music vs no music by headphones so that the investigator is blinded to the intervention. The outcome variable is amount of sedative used and self-reported anxiety level as reported on a 10 point visual analogue scale (VAS). The music intervention is begun 1 minute prior to the sedation procedure and continued until the subject is completely awake. Demographics will be collected for all patients. No identifiers are collected. Data will be compared for a change in VAS variable using non parametric methods.

DETAILED DESCRIPTION:
1. Objectives -The purpose of this study is to compare the amount of sedative (ketamine, propofol, ketofol, benzodiazepines, narcotics, or any other medications) used in procedural sedation of patients undergoing fracture reductions in the emergency department, as well as the amount of anxiety as measured by State-Trait Anxiety Inventory (STAI), in two groups: patients who listen to classical music during the procedure versus patients who do not listen to music during the procedure. The investigators hypothesize that patients who listen to classical music during procedural sedation will require lower amounts of sedatives and analgesia during the procedure and report lower levels of anxiety compared to patients who do not listen to classical music.
2. Background- Music has been used to reduce anxiety and the experience of pain during medical procedures and can reduce the requirements for sedation in particular procedures. One study looked at 100 patients who were undergoing interventional radiological procedures. After randomizing the participants in a 1:1 ratio, it was found that sedation was required in 42% of the patients in the music group compared to 60% of patients in the control group. Also, the mean dosage of midazolam was significantly less in the music group compared to the control group. This demonstrated a significant reduction in sedation requirements for patients who had self-selected music playing during interventional radiological procedures. Music effectively made the procedure safer by reducing the need for sedation and further contributed to the experience of the patient. Procedural sedation is used in the UNM Hospital (UNMH) Emergency Department (ED) on a regular basis to help patients tolerate orthopedic reductions of simple, closed fractures without needing to go through general anesthesia. This project is designed to use music therapy in an attempt to augment the effects of procedural sedation. Our investigation proposes to study whether music therapy as an adjunct to sedation decreases the amount of sedatives and analgesics used in orthopedic patients undergoing procedural sedation, and whether these patients report less anxiety by having music as an adjunct. Music therapy during procedures has been shown to be cost effective - it reduces patient sedation, procedural times, and number of staff members necessary to be present during procedures. Music therapy may also be effective in reducing anxiety in patients undergoing surgery with regional anesthesia: In a group of 80 patients assigned to an experimental and a control group, anxiety was significantly reduced in the experimental group who listened to music using headphones throughout the surgery. According to two systematic reviews, music therapy significantly improving pain scores, satisfaction scores, anxiety scores, heart rate, and arterial pressure.
3. Study-Wide Number of Subjects- Maximum target enrollment for each group will be 30 subjects, with a total of 60 subjects for project.
4. Study Timelines- In the experimental group, this music will be started 1 minute prior to conscious sedation and continued until the patient's sedation wears off and patient is again interactive with investigator. The study will take approximately 15 minutes of the patient's time, divided between time before the procedure and time after the procedure. The duration anticipated to enroll all study subjects is difficult to anticipate, as the UNMH ED receives as many as one conscious sedation patient a day and as few as one a week. However, the duration is anticipated to take less than two years. Once data collection has closed, it will take researchers no longer than one year to complete primary analysis.
5. Study Endpoints -The study endpoint will be reached when a total of 60 patients (30 experimental group and 30 in the control group) have been enrolled. There are no primary or secondary safety endpoints as there is no medical procedure or drug involved in this study.
6. Procedures Involved -Participants will be randomized into the intervention or control group. The intervention will be listening to a classical song. In the experimental group, this music will be started 1 minute prior to conscious sedation and continued until the patient's sedation wears off and patient is again interactive with investigator. The music will be played using an Apple™ IPOD player attached to headphones. During hours when study recruiters are available, all patients between 18-65 years of age presenting to the adult ED at UNMH and needing an orthopedic reduction with procedural sedation will be invited to participate. If a patient agrees to participate, a research associate will collect patient's background information (age, sex, type of fracture, location of fracture, etc.) and then administer the STAI scale. Subjects will be assigned to either the control or experimental group by flip of coin. Subjects will then undergo sedation and reduction, with research associate recording the doses of sedatives and analgesics used, at the times of push. Once patient returns to baseline, research associate will remove headphones and administer the STAI scale once again. Demographic information (age, sex, type of fracture, location of fracture, etc.), STAI scale scores, and the amount of sedatives and analgesics administered during the procedure. Please see data collection form attachment for a comprehensive list.
7. Provisions to Monitor the Data to Ensure the Safety of Subjects- The investigators are creating a Data and Safety Monitoring Plan for this study as the study is considered more than minimal risk by the investigational review board (IRB). The plan consists of monitoring the study for any adverse events incurred from subjects' participation in the study. Dr. Steven Weiss (also in Emergency Medicine) will head the management team. Every 6 months the investigators will evaluate the progress of the study, address any adverse events and create a report of any findings. At the yearly IRB renewal the investigator will include this report with the progress report. The endpoint will be when all subjects are recruited in the study, anticipated to take 18-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Any patient in the UNMH ED between age 18-65
* An upper extremity (defined as distal to humerus, including humerus) or lower extremity fracture (defined as distal to femur, including femur)
* A closed fracture
* Undergoing procedural sedation for reduction of the fracture in the emergency department.

Exclusion Criteria:

* Clinically intoxicated
* Have dementia
* Experiencing psychosis
* Are deaf
* Patient who do not speak English
* Adults unable to consent
* Pregnant women
* Prisoners will be excluded from participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Change in Visual analogue score | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Difference in STAI anxiety score before and after intervention | through study completion, an average of 1 year
Anxiety scale- pre and post | through study completion, an average of 1 year
Any positive finding on the Common Terminology Criteria for Adverse Events (CTCAEv4.0) psychiatric scale | through study completion, an average of 1 year
  Number of participants with treatment related adverse events as assessed by the 20 categories in the CTCAE v4.0 psychiatric scale.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ernst, MD, Principal Investigator — UNM hospital
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kulkarni S, Johnson PC, Kettles S, Kasthuri RS. Music during interventional radiological procedures, effect on sedation, pain and anxiety: a randomised controlled trial. Br J Radiol. 2012 Aug;85(1016):1059-63. doi: 10.1259/bjr/71897605. Epub 2012 Mar 14. PMID 22422386
- [Background] DeLoach Walworth D. Procedural-support music therapy in the healthcare setting: a cost-effectiveness analysis. J Pediatr Nurs. 2005 Aug;20(4):276-84. doi: 10.1016/j.pedn.2005.02.016. PMID 16030507
- [Background] Bae I, Lim HM, Hur MH, Lee M. Intra-operative music listening for anxiety, the BIS index, and the vital signs of patients undergoing regional anesthesia. Complement Ther Med. 2014 Apr;22(2):251-7. doi: 10.1016/j.ctim.2014.02.002. Epub 2014 Feb 23. PMID 24731896
- [Background] Wang MC, Zhang LY, Zhang YL, Zhang YW, Xu XD, Zhang YC. Effect of music in endoscopy procedures: systematic review and meta-analysis of randomized controlled trials. Pain Med. 2014 Oct;15(10):1786-94. doi: 10.1111/pme.12514. Epub 2014 Aug 19. PMID 25139786
- [Background] Yinger OS, Gooding LF. A systematic review of music-based interventions for procedural support. J Music Ther. 2015 Spring;52(1):1-77. doi: 10.1093/jmt/thv004. Epub 2015 Apr 15. PMID 25878063